CLINICAL TRIAL: NCT07143682
Title: Letrozole Step up Compared to Conventional Protocol for Ovulation Induction in Infertile Women With Polycystic Ovary Syndrome
Brief Title: Letrozole Step up Protocol for Ovulation Induction in Infertile Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Shakeela Ishrat, Professor Shakeela Ishrat, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4286
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Infertility
Keywords: Polycystic ovary syndrome; letrozole; ovulation induction
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Congresses as Topic; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole step up (Experimental): Tab letrozole 2.5mg one, two, three, and four tablets once daily from 2nd/3rd day of the menstrual cycle for 4 days
  Interventions: Drug: Letrozol step up dose
- Conventional fixed dose letrozole (Active Comparator): Tab letrozole 5mg once daily for 5 days started from the 2nd/3rd day of the menstrual cycle
  Interventions: Drug: Conventional fixed dose letrozole

INTERVENTIONS:
Drug: Letrozol step up dose — Tablet letrozole 2.5mg one, two, three, and four tablets once daily from 2nd/3rd day of the menstrual cycle for 4 days
  Arms: Letrozole step up
Drug: Conventional fixed dose letrozole — Tab letrozole 5mg once daily for 5 days started from the 2nd/3rd day of the menstrual cycle
  Arms: Conventional fixed dose letrozole

SUMMARY:
The goal of this clinical trial is to learn if drug letrozole in step up dose works better to treat anovulation in infertile women with polycystic ovary syndrome. It will also learn about the safety of drug letrozole in step up dose. The main Questions it aims to answer are:

* Does drug letrozole in step up dose result in better ovarian response?
* What medical problems do participants have when taking drug letrozole in step up dose? Researchers will compare drug letrozole step up dose to a standard low dose to see if the step up dose works to achieve better ovarian response.

Participants will:

* Take drug letrozole step up or standard low dose from day 2 of menstruation for 3 cycles
* Visit the clinic on day 12-16 of menstural cycle for checkups and tests
* Keep a diary of any untoward symptoms

DETAILED DESCRIPTION:
Background: Polycystic ovary syndrome (PCOS) is the largest single cause of anovulatory infertility. Letrozole, an aromatase inhibitor, has been regarded as the first-line drug for ovulation induction in PCOS patients. The conventional protocol of letrozole includes the administration of a fixed dose of letrozole (2.5 -7.5 mg) for 5 days. Few recent studies have shown that the step-up letrozole protocol causes more follicles to grow, induces more ovulation, and increases the pregnancy rate. This study aimed to compare the effect of the letrozole step-up and conventional fixed-dose protocol for ovulation induction in infertile women with PCOS.

Methods: This open-label randomized controlled study was conducted on a total of 70 infertile PCOS women eligible for ovulation induction. Treatment with letrozole started from day 2-3 of menstruation or withdrawal bleeding. They were randomly allocated into two groups. The experimental group (n=35) was given step-up letrozole, one (2.5 mg), two (5 mg), three (7.5 mg), and four (10 mg) tablets, single dose sequentially for 4 days. The comparator group (n=35) received conventional fixed-dose letrozole, two (5mg) tablets daily for 5 days. The outcome variables were the number of participants having a mature follicle by day 12-16 of the cycle and the number of mature follicles on the day of trigger.

ELIGIBILITY:
Inclusion Criteria:

* PCOS women with subfertility
* Selected for ovulation induction

Exclusion Criteria:

* Body mass index (BMI) ˂18 and ≥30 kg/m2,
* Women with other infertility factors (endometriosis, suspected tubal factor, and uterine causes of infertility)
* Male factor infertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The number of participants having mature follicle (mean diameter ≥18mm) | 3 months
  The number of participants having mature follicle (mean diameter ≥18mm) on day 12 to 16 of the cycle
The number of participants having adequate endometrial thickness ( 7mm or more) | 3 months
  The number of participants having adequate endometrial thickness ( 7mm or more) on the day of trigger

SECONDARY OUTCOMES:
Pregnancy | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaur J, Suri V, Gainder S, Arora A. Prospective randomized trial comparing efficacy of letrozole step-up protocol with letrozole plus gonadotropins for controlled ovarian stimulation and intrauterine insemination in patients with unexplained infertility. Arch Gynecol Obstet. 2019 Dec;300(6):1767-1771. doi: 10.1007/s00404-019-05326-2. Epub 2019 Oct 20. PMID 31631248